CLINICAL TRIAL: NCT05323890
Title: Neoadjuvant Tislelizumab Combined With Chemoradiotherapy for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma : Single Arm Phase II Study
Brief Title: Tislelizumab Combined With Neoadjuvant Radiotherapy and Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Xue Meng, Ph.D, M.D, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shandong CHI
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Advanced Esophageal Squamous Cell Cancer
MeSH Terms: interventions — Neoadjuvant Therapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tislelizumab arm (Experimental): Radiotherapy: PTV 41.4Gy in 23 Fractions，5 days per week; Chemotherapy: Paclitaxel (Albumin bound) (100mg/m2) and Cisplatin (75 mg/m2) for 5 weeks, concurrent with radiotherapy; Immunotherapy: Tislelizumab (200mg per 3 weeks)
  Interventions: Drug: Tislelizumab Combined With Neoadjuvant Radiotherapy and Chemotherapy

INTERVENTIONS:
Drug: Tislelizumab Combined With Neoadjuvant Radiotherapy and Chemotherapy — Patients received tislelizumab at a fixed dose of 200 mg every three weeks (q3w, 21 days) for 2 cycles.
  Other Names: Anti-PD-1 Therapy

SUMMARY:
This study aimed to evaluate the safety and feasibility of neoadjuvant tislelizumab combined with chemoradiotherapy in patients with resectable esophageal squamous cell cancer. The tumor microenvironment and circulating immunological biomarkers in these patients were further evaluated to explore the factors affecting the efficacy of neoadjuvant therapy for esophageal cancer. This study will provide valuable information for further prospective clinical trials of neoadjuvant anti-PD-1 and other immunotherapy in esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Histologically or cytologically confirmed resectable squamous-cell esophageal cancer ( cT1-2N+/ cT3-4aN0-3M0)
3. Eastern Cooperative Oncology Group (ECOG) status 0-1
4. Signed written informed consent prior to the implementation of any trial-related rocedures
5. Adequate organ function, evidenced by laboratory results with no contraindications to chemotherapy Absolute neutrophil count ≥ 1,500 х109/l Thrombocytes ≥ 100 х 109/l Hemoglobin ≥ 90 mg/l Creatinine ≤ 1.5 x ULN or creatinine clearance (calculated using the Cockcroft-Gault formula) ≥40 mL/min Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN) Alkaline phosphatase (ALP) > 5 x ULN Bilirubin > 1.5 х ULN

Exclusion Criteria:

1. Patients diagnosed with any other malignant tumor
2. Patients at risk for tracheoesophageal fistula or aortoesophageal fistula
3. Have received prior therapy with: chemotherapy, radiation therapy,immune checkpoint inhibitor
4. Insufficient caloric and/or fluid intake despite consultation with a dietitian and/or tube feeding
5. Have an active infection requiring systemic therapy that has not resolved 3 days (simple infection, such as cystitis) to 7 days (severe infection, such as pyelonephritis) before the first dose of trial treatment
6. Patients who cannot tolerate chemoradiotherapy or surgery due to severe cardiac, lung dysfunction
7. A history of interstitial lung disease or non-infectious pneumonia
8. Active autoimmune disease with systemic therapy (ie, use of disease modifiers, corticosteroids, or immunosuppressive drugs) in the past 2 years
9. Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibody) and various viral hepatitis infections
10. Patients who have received allogeneic stem cell or solid organ transplantation
11. Women during pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response Rate | From date of surgery to 14 days later
  No more than 10% of tumor cells were found in neoadjuvant surgical specimens.
Pathologic complete response rate | From date of surgery to 14 days later
  Pathologic complete response rate

SECONDARY OUTCOMES:
Disease free survival | 24 months
  Disease free survival will be calculated from the start of the treatment to the disease progression or death of any reason.
Incidence of Treatment-related Adverse Events | 8 weeks
  Number and percentage of cases of all adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China